CLINICAL TRIAL: NCT05325177
Title: A Pilot, Randomized Controlled Study of the Effects of High Dose Ibuprofen on Cerebral and Splanchnic Tissue Oxygenation During Treatment of Hemodynamically Significant Patent Ductus Arteriosus (hsPDA) in Preterm Infants
Brief Title: PDA Treatment With Ibuprofen and Changes in Tissue Oxygenation.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NICU-PDA-01
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
Keywords: Ibuprofen
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: The investigators are equipped with unique and complementary expertise that will propel this promising work forward. We will recruit 30 preterm infants less than (<)29 weeks gestation at birth with echocardiographic evidence of hsPDA that require pharmacologic treatment. We will examine renal, cerebral, intestinal blood flow and tissue oxygenation in high-risk preterm infants receiving high dose or standard-dose Ibuprofen treatment for hsPDA. Successful completion of this study will establish feasibility and provide proof-of-concept for a future multi-center trial. We will use descriptive statistics to compare patients' characteristics. To compare NIRS and Doppler data between the two groups, we will use paired t-test if data is normally distributed or Wilcoxon signed-rank test if not normally distributed
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 infants (Active Comparator): (n=15) will receive three doses of standard-dose Ibuprofen. (10-5-5 mg/kg) 1 dose every 24 hours after enrollment, for a total of 3 doses
  Interventions: Drug: Standard Dose Ibuprofen
- Group 2 infants (Active Comparator): (n = 15) will receive three doses of high-dose Ibuprofen Motrin. (20-10-10 mg/kg) 1 dose every 24 hours after enrollment, for a total of 3 doses
  Interventions: Drug: High Dose Ibuprofen

INTERVENTIONS:
Drug: Standard Dose Ibuprofen — (10-5-5 mg/kg) 1 dose every 24 hours after enrollment, for a total of 3 doses
  Arms: Group 1 infants
Drug: High Dose Ibuprofen — (20-10-10 mg/kg) 1 dose every 24 hours after enrollment, for a total of 3 doses
  Arms: Group 2 infants

SUMMARY:
Babies who are born very prematurely are often born with murmurs in the heart. In preterm babies, one of the most common causes of murmur is the presence of a PDA. This is the persistence of a connection that normally exists in the baby before it is born, connecting between the major blood vessels that leave the heart. In term babies, this channel closes shortly after birth when normal adult circulation is achieved. However, in preterm babies, the PDA can remain open, which can lead to multiple problems in the baby.

Our current standard of treatment in the Neonatal Intensive Care Unit (NICU) is to perform cardiac ultrasound (echocardiogram) in all babies less than 29 weeks gestation to diagnose the presence of hsPDA. We also use an echocardiogram to follow the PDA until complete closure. If present, the standard treatment in the NICU is to give medication, usually Ibuprofen, a non-steroidal anti-inflammatory drugs (NSAID), to close the PDA.

Near-infrared spectroscopy (NIRS) is a new type of device to detect oxygenated blood supply to the brain, kidney, and abdominal regions. This device is used to assess the effects of Ibuprofen on oxygen supply to these three regions.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than (< )29 weeks gestation at birth
* Echocardiographic evidence of hsPDA (as outlined in the NICU PDA treatment guidelines) at 7-21 days of life requiring pharmacologic treatment as determined by the managing physician.

Exclusion Criteria:

* Not able to consent for any reason
* Preterm infants with congenital heart disease except for PDA, PFO (patent foramen ovale), small and restrictive ASD (atrial septal defect), or small VSD (ventricular septal defect).
* Preterm infants with lethal genetic malformations.
* Preterm infants with congenital abdominal wall defects (omphalocele, gastroschisis).
* Preterm infants with congenital or acquired brain anomaly.
* Infants who receive ibuprofen for PDA treatment during the first week of life will be excluded. We will recruit infants between day 7 and 21 only because high-dose ibuprofen is not indicated during the first week of life
* Preterm infants with contraindications to Ibuprofen therapy, including severe intraventricular hemorrhage (IVH), low platelet count < 50,000 platelets per microliter, renal impairment with creatinine >160 mmol/L or necrotizing enterocolitis (NEC) > Stage 2 (using modified bell's Criteria).
* Preterm infants with spontaneous intestinal perforation (SIP).
* Acute kidney injury (defined as an increase in serum creatinine of 50% or more from the previous lowest value or a urinary output of less than 1 mL/kg per hr.).

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in regional tissue oxygenation (splanchnic, cerebral, and the splanchnic-cerebral oxygenation ratio 'SCOR') during hsPDA treatment | with the first 28 days after enrolment
Change in splanchnic, cerebral, and renal Doppler blood flow during hsPDA treatment [Peak Systolic Velocity (PSV), End Diastolic Velocity (EDV), and Resistive Index (RI)] | with the first 28 days after enrolment

SECONDARY OUTCOMES:
Necrotizing Enterocolitis (NEC): > 2 (Modified bell's Criteria) | with the first 28 days after enrolment
Spontaneous intestinal perforation (SIP) | with the first 28 days after enrolment
Incidence of oliguria | (<1 ml/kg/hour for > 12 hours)
Feeding intolerance | with the first 28 days after enrolment
  we define feeding intolerance as the decision by the managing team to withhold feeds for at least 24 hours in the absence of definite evidence of medical or surgical NEC
Gastrointestinal bleeding | with the first 28 days after enrolment
  Any amount of visible bright red or altered blood in emesis, nasogastric tube, or feces
Pulmonary hemorrhage | with the first 28 days after enrolment
Presence of echocardiographic features of pulmonary hypertension | with the first 28 days after enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa General Hospital, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No